CLINICAL TRIAL: NCT00939198
Title: Determination of Prevalence and Intensity of Hookworm Infection and Community Preparedness for Hookworm Vaccine Trials in Endemic Areas of Northeastern Minas Gerais, Brazil
Brief Title: Prevalence of Hookworm Infection and Community Preparedness for Hookworm Vaccine Trials in Endemic Areas of Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert B. Sabin Vaccine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SVI-06-01
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Hookworm Infection
Keywords: Hookworm; Allergy; Vaccine; Skin Test; Immediate-type hypersensitivity to Na-ASP-2 hookworm antigen
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Na-ASP-2 Hookworm Antigen Skin Test (Experimental): All participants will be skin tested with Na-ASP-2 skin test reagent applied to their arms, using both the prick-puncture and intradermal techniques.
  Interventions: Biological: Na-ASP-2 Skin Test Reagent

INTERVENTIONS:
Biological: Na-ASP-2 Skin Test Reagent — Na-ASP-2 Hookworm Skin Test Reagent, 1-1000 mcg/mL solution

SUMMARY:
Na-ASP-2 is a protein expressed during the larval stage of the N. americanus hookworm life cycle. In a clinical study in previously hookworm-infected adults in Brazil, this protein induced urticarial reactions (rash) in a subset of volunteers. The clinical trial component of this study involves skin testing for immediate-type hypersensitivity to the Na-ASP-2 Antigen. Both prick-puncture and intradermal tests will be applied.

DETAILED DESCRIPTION:
The clinical testing of the Na-ASP-2 Skin Test Reagent to detect Immediate-type hypersensitivity to the Na-ASP-2 hookworm antigen will be conducted as part of a larger, on-going observational study of the prevalence and intensity of hookworm infection currently underway in Brazil. Eligible adult participants (ages 18-45 years) in this observational study will be invited to undergo the skin testing procedure. Skin testing will only be performed if they agree and sign the supplemental informed consent form for this skin testing procedure.

* Study site: Americaninhas Vaccine Center, Americaninhas, Minas Gerais, Brazil
* Number of participants to be skin tested: approximately 150 adults
* Duration of the skin testing procedures: up to 1 month; each participant will undergo skin testing and a follow-up blood collection 21+/-7 days after skin testing.
* Each participant will have both skin prick-puncture and intradermal skin tests applied on the same study day. The prick-puncture and intradermal tests will be applied sequentially to the volar aspects of the participant's forearms:

  1. Skin prick-puncture: three different concentrations of Na-ASP-2 solution (10, 100, and 1000 μg/mL) will be applied sequentially in duplicate, to the left forearm.
  2. Intradermal: one concentration of Na-ASP-2 (100 μg/mL) will be injected, in duplicate, to the right forearm.
  3. Allergen diluent and histamine solutions will be utilized as the negative and positive controls, respectively, for both the skin prick-puncture and intradermal tests.
  4. Participants will be observed in the study clinic for at least 30 minutes following application of the skin tests, and will be examined 2 and 7 days following skin testing.
  5. Sizes of the wheal and erythema reactions for each application will be recorded and graded in comparison to the histamine positive control reaction.
* Each participant will have blood collected via venipuncture (a maximum of 25 mL) immediately prior to application of the skin tests, and between 2 and 4 weeks after skin testing, in order to measure antibodies (particularly IgG and IgE) to Na-ASP-2 using an ELISA procedure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 6 and 45 years of age, inclusive, at the time of consenting to the parent study.
* Age greater than or equal to 18 years at the time of signing the supplemental informed consent document for the skin test procedure (parent study).
* Willingness to participate in the study as evidenced by signing the informed consent or assent document.

Exclusion Criteria:

* Inability to correctly answer all questions on the informed consent comprehension questionnaire.
* Attends school or works full-time outside of the study area.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer to participate in the trial or would render the subject unable to comply with the protocol.
* Pregnancy as determined by a positive urine hCG test (if female).
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of planned skin test application.
* Extensive dermatitis precluding skin testing.
* Current use of a beta blocker (oral or topical) or anti-histamine medication. A volunteer may participate in the study if they agree to withhold use of an anti-histamine for at least 5 days prior to application of the skin test.
* Use of a tricyclic anti-depressant within the past month.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bethony, PhD, Principal Investigator — Albert B. Sabin Vaccine Institute
Locations (1):
- Centro de Pesquisas Rene Rachou, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Fujiwara RT, Bethony J, Bueno LL, Wang Y, Ahn SY, Samuel A, Bottazzi ME, Hotez P, Mendez S. Immunogenicity of the hookworm Na-ASP-2 vaccine candidate: characterization of humoral and cellular responses after vaccination in the Sprague Dawley rat. Hum Vaccin. 2005 May-Jun;1(3):123-8. doi: 10.4161/hv.1.3.1924. Epub 2005 May 20. PMID 17012856
- [Background] Goud GN, Bottazzi ME, Zhan B, Mendez S, Deumic V, Plieskatt J, Liu S, Wang Y, Bueno L, Fujiwara R, Samuel A, Ahn SY, Solanki M, Asojo OA, Wang J, Bethony JM, Loukas A, Roy M, Hotez PJ. Expression of the Necator americanus hookworm larval antigen Na-ASP-2 in Pichia pastoris and purification of the recombinant protein for use in human clinical trials. Vaccine. 2005 Sep 15;23(39):4754-64. doi: 10.1016/j.vaccine.2005.04.040. PMID 16054275
- [Background] Diemert DJ, Bethony JM, Hotez PJ. Hookworm vaccines. Clin Infect Dis. 2008 Jan 15;46(2):282-8. doi: 10.1086/524070. PMID 18171264

RESULTS

PARTICIPANT FLOW:
Groups:
- Na-ASP-2 Hookworm Antigen Skin Test: All participants will be skin tested with Na-ASP-2 skin test reagent (1000 mcg/ml recombinant Na-ASP-2) applied to their arms, using both the prick-puncture and intradermal techniques.
Period: Overall Study
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Started | 87
Completed | 87
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Number analyzed (Participants) | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 87
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 87
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 87

OUTCOME MEASURES:

1. Primary Outcome: Size of Wheal Diameter at Site of Skin Test Application, Measured 15 Minutes After Injection
Time Frame: 15 minutes after skin test application
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Number analyzed (Participants) | 87
cm | 3.5 [0 to 6.5]

2. Secondary Outcome: Anti-Na-ASP-2 IgE Antibody Level on Day of Skin Test Reaction
Time Frame: Upon skin testing
Measure: Median (Inter-Quartile Range); unit: kU/L
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Number analyzed (Participants) | 42
kU/L | 1.89 [0.36 to 5.11]

ADVERSE EVENTS:
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Serious Adverse Events (participants affected / at risk) | 0/87
Other Adverse Events (participants affected / at risk) | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No